CLINICAL TRIAL: NCT04067570
Title: Post-Prostatectomy Linac-Based Ultrahypofractionated Radiotherapy for Patients With Localized Prostate Cancer: A Treatment Feasibility and Outcomes Study
Brief Title: Post-Prostatectomy Linac-Based Ultrahypofractionated Radiotherapy for Patients With Localized Prostate Cancer
Acronym: PLUTO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Chia-Lin (Eric) Tseng, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLUTO
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: SBRT; Radical Prostatectomy
Keywords: Prostate cancer; Radiation; Ultrahypofractionated Radiotherapy; PSA Rise; SBRT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT post operative (Experimental): Stereotactic Body Radiotherapy (SBRT) 30 Gy in 5 fractions, once weekly to prostate bed
  * / - 25 Gy in 5 fractions, once weekly simultaneously to pelvic lymph nodes
  * / - 6-24 months of androgen deprivation therapy (ADT)
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Stereotactic body radiation therapy, or SBRT, is a cancer treatment that delivers extremely precise, very intense doses of radiation to cancer cells while minimizing damage to healthy tissue

SUMMARY:
Radical prostatectomy is a common treatment for localized prostate cancer. More than 30% of men who undergo surgery will subsequently develop recurrence, particularly in patients with adverse features where the risk may be even higher. Recurrence typically manifests as a rise in serum-level of prostate-specific antigen (PSA), referred to as biochemical recurrence. Post-operative radiotherapy is a potentially curative option for many patients, as shown in multiple prior randomized studies. A standard course of post-operative radiation requires 6 to 6 and half weeks of treatment, 5 days a week; however, new high-precision radiation techniques with image guidance, termed stereotactic body radiotherapy (SBRT), can deliver an equivalent or higher dose of treatment in 5 visits. Our group, amongst others, have demonstrated in previous studies, that the new 5-treatment technique was safe, convenient and effective in patients with intact prostates. Currently, limited data exists on this approach after prostatectomy. This study will be one of the first to assess the side effect profile and efficacy of SBRT in patients with localized prostate cancer who are considered candidates for post-prostatectomy radiation.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed diagnosis of adenocarcinoma of the prostate

  * Completed written informed consent
  * Able and willing to complete self report questionnaires
  * Pathologic stage T3 or T4 (without any gross residual disease), NX-0, M0, and/or +ve surgical margins, and/or a rising PSA post-radical prostatectomy on at least 2 consecutive measurements

Exclusion Criteria:

* • Gross residual disease

  * Histological or radiological node +ve (N1) or distant metastases (M1)
  * Prior pelvic radiotherapy
  * Contraindications to radical pelvic radiotherapy (e.g. connective tissue disease or inflammatory bowel disease)
  * Hip prosthesis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Prostate Cancer- male patients only
Enrollment: 30 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Acute genitourinary (GU) and gastrointestinal (GI) toxicities | Through accrual completion, up to 3 years
  Based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Incidence of late GU and GI toxicities (≥6 months) | Through accrual completion, up to 3 years
  Using CTCAE v5.0
Biochemical disease-free survival (bDFS) | Through study completion, up to 3 years
  Biochemical disease-free survival (bDFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided